CLINICAL TRIAL: NCT00187317
Title: Development and Evaluation of a Perturbation-based Balance-training Program for Older Adults
Brief Title: Evaluation of a Balance-recovery Specific Falls Prevention Exercise Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Brian Maki, Centre for Studies in Aging
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NET-54025-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Accidental Falls
Keywords: Exercise; Rehabilitation; Postural Balance; Accidental Falls; Geriatrics
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Pliability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PERT (Experimental): Perturbation-based balance training.
  Interventions: Behavioral: Balance training (exercise)
- CON (Placebo Comparator): Flexibility and relaxation training.
  Interventions: Other: Flexibility and relaxation exercise

INTERVENTIONS:
Behavioral: Balance training (exercise) — Perturbation-based balance training. 30-minute sessions three times per week for six weeks.
  Arms: PERT
Other: Flexibility and relaxation exercise — 30-minute sessions, three times per week for six weeks.
  Arms: CON

SUMMARY:
This study aims to investigate the potential to train compensatory stepping and grasping reactions for the prevention of falls.

DETAILED DESCRIPTION:
Physical activity and exercise have been shown to prevent falling in older adults, although the exact mechanisms by which exercise prevents falls is unclear. Compensatory stepping and grasping reactions are frequently used to prevent a fall to the ground following a loss of balance. Age-related impairment in these reactions may be related to an increased risk of falling. Therefore, the purpose of this study is to investigate means for reversing age-related impairment in compensatory stepping and grasping reactions. A training program involving perturbation-evoked reactions will be evaluated.

Comparison(s): Balance recovery ability before and after a 6-week training program will be assessed. Performance of the training group will be compared to a control group not receiving stepping and grasping training.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling
* History of falls (at least 1 fall in the past 12 months) or poor balance
* Functional mobility (no dependence on mobility aids)

Exclusion Criteria:

* Neurological or musculoskeletal disorder
* Cognitive disorder (e.g. dementia)
* Osteoporosis

Ages: 64 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-11; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Ability to recover balance by stepping and grasping | Before and after 6-week intervention

SECONDARY OUTCOMES:
Fall frequency; clinical measures related to balance and fall risk (e.g. FallScreen, Community Balance and Mobility Scale, balance confidence) | One year post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brian Maki, PhD, PEng, Principal Investigator — Sunnybrook & Women's College Health Sciences Centre; University of Toronto
Locations (1):
- Centre for Studies in Aging, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Maki BE, McIlroy WE, Perry SD. Influence of lateral destabilization on compensatory stepping responses. J Biomech. 1996 Mar;29(3):343-53. doi: 10.1016/0021-9290(95)00053-4. PMID 8850640
- [Background] Province MA, Hadley EC, Hornbrook MC, Lipsitz LA, Miller JP, Mulrow CD, Ory MG, Sattin RW, Tinetti ME, Wolf SL. The effects of exercise on falls in elderly patients. A preplanned meta-analysis of the FICSIT Trials. Frailty and Injuries: Cooperative Studies of Intervention Techniques. JAMA. 1995 May 3;273(17):1341-7. PMID 7715058
- [Background] Rogers MW, Johnson ME, Martinez KM, Mille ML, Hedman LD. Step training improves the speed of voluntary step initiation in aging. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):46-51. doi: 10.1093/gerona/58.1.m46. PMID 12560410
- [Background] McIlroy WE, Maki BE. Age-related changes in compensatory stepping in response to unpredictable perturbations. J Gerontol A Biol Sci Med Sci. 1996 Nov;51(6):M289-96. doi: 10.1093/gerona/51a.6.m289. PMID 8914501
- [Background] Maki BE, McIlroy WE. Change-in-support balance reactions in older persons: an emerging research area of clinical importance. Neurol Clin. 2005 Aug;23(3):751-83, vi-vii. doi: 10.1016/j.ncl.2005.01.002. No abstract available. PMID 16026675
- [Background] Maki BE, Cheng KC, Mansfield A, Scovil CY, Perry SD, Peters AL, McKay S, Lee T, Marquis A, Corbeil P, Fernie GR, Liu B, McIlroy WE. Preventing falls in older adults: new interventions to promote more effective change-in-support balance reactions. J Electromyogr Kinesiol. 2008 Apr;18(2):243-54. doi: 10.1016/j.jelekin.2007.06.005. Epub 2007 Sep 4. PMID 17766146
- [Result] Mansfield A, Peters AL, Liu BA, Maki BE. A perturbation-based balance training program for older adults: study protocol for a randomised controlled trial. BMC Geriatr. 2007 May 31;7:12. doi: 10.1186/1471-2318-7-12. PMID 17540020
- [Result] Mansfield A, Peters AL, Liu BA, Maki BE. Effect of a perturbation-based balance training program on compensatory stepping and grasping reactions in older adults: a randomized controlled trial. Phys Ther. 2010 Apr;90(4):476-91. doi: 10.2522/ptj.20090070. Epub 2010 Feb 18. PMID 20167644